CLINICAL TRIAL: NCT04620317
Title: Effects of Synbiotics on Functional Constipation and Other Contributing Factors Among Constipated Individuals in Serdang, Selangor, Malaysia
Brief Title: Effects of Synbiotics on FC and Other Contributing Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr. Rosita Jamaluddin, Assoc. Prof. Dr., Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SynFC_001
Record Dates: First submitted 2018-10-16; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Functional Constipation
Keywords: Prevalence; functional constipation; Rome III criteria; Bristol Stool Form Scale; defecation frequency; PAC-SYM; PAC-QOL; randomised controlled trial (RCT); synbiotic
MeSH Terms: interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic (Active Comparator): The product contained three clinically studied active ingredients namely inulin-oligofructose (prebiotic; derived from chicory root), at least 6 billion (B) colony forming unit (CFU) of Lactobacillus plantarum LP01 (probiotic) and 4 B CFU of Bifidobacterium lactis BB12 (probiotic) per sachet.
  Interventions: Dietary Supplement: Synbiotic
- Placebo (Placebo Comparator): Placebo contains only maltodextrin without any active ingredients, equally same in physical form, freeze-dried white powder with characteristic odor and water soluble as the synbiotic supplement.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic — 10 billion (B) colony forming unit (CFU) of Lactobacillus plantarum LP01, Bifidobacterium lactis BB12, and inulin oligofructose
  Arms: Synbiotic
Dietary Supplement: Placebo — Non-active ingredients - Maltodextrins
  Arms: Placebo

SUMMARY:
Prevalence of functional constipation (FC) was first determined with 15.2% reported. Next, a 16-week randomised, double-blind, placebo-controlled study conducted to assess the improvement in functional constipation among the respective individuals by using synbiotic supplement. Throughout the intervention, it was reported that significant improvements for defecation frequency, Bristol Stool Form (BSF) scale, and Patients Assessment of Constipation Symptoms (PAC-SYM) scores were reported within synbiotic group (p < 0.001). However, no significant different was reported when compared both groups as placebo group was found to have significant within-group difference too. Placebo effect was suspected in this study.

DETAILED DESCRIPTION:
Digestive system disease is the top ten principal causes of morbidity and mortality among Malaysians whereby functional constipation (FC) is the commonest functional gastrointestinal disorders (FGIDs) reported. Although numerous treatments are available, but over-the-counter drugs which have low product safety and possible toxicity were always given as the treatment option. Synbiotic have been well-studied to improve digestive health includes constipation. Thus, the objectives of this study were to determine the prevalence of FC and to evaluate the effects of synbiotic supplement on improving FC symptoms and contributing factors among constipated individuals in Serdang, Selangor. This study comprised of two parts which were screening and intervention part. The prevalence of functional constipation was relatively high in the study community. Synbiotic supplement was effective in the improvement of functional constipation symptoms, quality of life, and psychological factors. However, the positive improvement in placebo group indicated the existence of placebo effects which led to the improvement in quality of life and changes in psychological factors. Therefore, the current findings are useful information for future intervention in improving functional constipation symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian of either gender;
* 18 to 65 years old;
* Body mass index (BMI) 16.0 to 29.9 kg/m2;
* Positively diagnosed with functional constipation with Rome III-defined constipation module by the gastroenterologist

Exclusion Criteria:

* Vulnerable groups of pregnant and breastfeeding women;
* Physically or mentally handicapped individuals;
* Diagnosed with organic constipation (constipation associated with any neoplastic diseases, neuropathy or mechanical obstruction);
* Diagnosed with cardiovascular diseases, diabetes mellitus, cancer, neurological disease or other serious illnesses or severe medical complications;
* Faced alarm features indicative of colorectal cancer, metabolic disease and a history of gastrointestinal surgery.

To avoid the likelihood of co-intervention bias, the following respondents were excluded:

* On gastrointestinal medications;
* Consumed probiotics or synbiotic products more than once a week in two weeks preceding screening or during intervention period;
* Regularly used laxatives (more than once per week), used anticholinergics, anti-diarrheals, antibiotics or laxative in two weeks preceding screening or at any point during intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Defecation frequency | 16 weeks
  Defecation frequency was measured through participants' self reported defecation frequency in a week.
Stool types - Bristol Stool Form (BSF) Scale | 16 weeks
  BSF scale was used to characterise human stools to seven classifications using seven pictorial presentation of stool types.Type 1 stool shows the very slow transit time with longest time spent in the colon whereas Type 7 indicates the least time spent in the colon and has fast bowel transit time. Meanwhile, Type 4 is the most ideal stool type optimal colonic transit time.
Constipation symptoms - Patients Assessment of Constipation Symptoms (PAC-SYM) | 16 weeks
  PAC-SYM consists of a total of 12 questions includes abdominal symptoms, rectal symptoms, and stool symptoms. It comprised with a 5-point Likert scale ranging from 0 (Absent) to 4 (Very severe). The values of subscales and total scores for PAC-SYM were then computed as average item response within the scales and for the global score. Lower score obtained indicates less symptom severity.

SECONDARY OUTCOMES:
Quality of life - Patients Assessment of Constipation Quality of Life (PAC-QOL) | 16 weeks
  Quality of life was measured using Patients Assessment of Constipation Quality of Life (PAC-QOL). PAC-QOL consists of a total of 28 questions which was grouped into four domains include physical discomfort, psychological discomfort, worries and concerns, and satisfaction. It comprised with a 5-point Likert scale ranging from 0 (Not at all/None of the time) to 4 (Extremel/All of the time).The values of subscales and total scores for PAC-QOL scores were then computed as average item response within the scales and for the global score. Lower score point indicates a better quality of life of the respective participant.
Psychological factor - Depression, Anxiety, and Stress scale (DASS) | 16 weeks
  Psychological factor was measured using Depression, Anxiety, and Stress scale (DASS). DASS was used to self-report the severity of depression, anxiety and stress level. The questionnaire based on 4-point Likert scale, ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much, or most of the time). The scores of depression, anxiety, and stress were summated for the relevant items followed by categorised to the severity of the condition. Lower score point indicates a less severity of the respective participant.